CLINICAL TRIAL: NCT04141072
Title: Shrunken Pore Syndrome's Effect on Mortality in Elective Cardiac Surgery
Brief Title: Shrunken Pore Syndrome: a Retrospective, Single Center, Cohort Study
Status: Completed | Type: Observational
Sponsor: Henrik Bjursten (Other)
Responsible Party: Sponsor-Investigator, Henrik Bjursten, Assoc. Prof, Region Skane
Organization: Region Skane (Other)
Other Study IDs: SPS
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Kidney Diseases
Keywords: CKD; Creatinine; Cystatin C; Cardiac surgery; GFR
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

INTERVENTIONS:
Diagnostic Test: Shrunken Pore Syndrome — eGFR Cystatin C ≤ 60% of eGFR Creatinine

SUMMARY:
To study the impact a difference in renal clearance of small and large molecules has on long-term survival.

DETAILED DESCRIPTION:
Renal dysfunction is considered a major risk factor in cardiac surgery. Renal function has earlier been estimated by creatinine and more recently by cystatin C, both of which are analysed in a blood sample. New evidence seems to suggest that if the ratio between estimated renal function from cystatin C and creatinine is below 60% the patient has a higher rate of mortality irrespective of renal function. This syndrome is named Shrunken Pore Syndrome.

We study patients whom have undergone elective cardiac surgery at our institution and on whom we before the surgery has collected blood samples. They are all included in our in house patient registry and qulaity database and afterwards we match this data to our national tax registry to get data on mortality.

Our aim is to evaluate whether Shrunken Pore Syndrome influence mortality following elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG and/or sAVR at the department of Cardiothoracic Surgery, Skåne University Hospital in Lund, Sweden between 1 January 2010 and 31 December 2015.

Exclusion Criteria:

* Emergency operation
* Redo operation
* Preoperatively missing cystatin C or creatinine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skåne University Hospital in Lund is a tertiary care hospital that is the sole provider of cardiac surgery to the Southern part of Sweden, comprising 1 500 000 people.
Sampling Method: Probability Sample
Enrollment: 4719 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Mortality during follow up | 1 January 2010 - 1 January 2019
  All cause mortality at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Bjursten, MD PhD, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dardashti A, Nozohoor S, Grubb A, Bjursten H. Shrunken Pore Syndrome is associated with a sharp rise in mortality in patients undergoing elective coronary artery bypass grafting. Scand J Clin Lab Invest. 2016;76(1):74-81. doi: 10.3109/00365513.2015.1099724. PMID 26647957
- [Background] Grubb A, Lindstrom V, Jonsson M, Back SE, Ahlund T, Rippe B, Christensson A. Reduction in glomerular pore size is not restricted to pregnant women. Evidence for a new syndrome: 'Shrunken pore syndrome'. Scand J Clin Lab Invest. 2015 Jul;75(4):333-40. doi: 10.3109/00365513.2015.1025427. PMID 25919022
- [Result] Herou E, Dardashti A, Nozohoor S, Zindovic I, Ederoth P, Grubb A, Bjursten H. The mortality increase in cardiac surgery patients associated with shrunken pore syndrome correlates with the eGFRcystatin C/eGFRcreatinine-ratio. Scand J Clin Lab Invest. 2019 May;79(3):167-173. doi: 10.1080/00365513.2019.1576101. Epub 2019 Feb 15. PMID 30767571
- [Derived] Herou E, Grubb A, Dardashti A, Nozohoor S, Zindovic I, Ederoth P, Bjursten H. Reduced renal elimination of larger molecules is a strong predictor for mortality. Sci Rep. 2022 Oct 20;12(1):17517. doi: 10.1038/s41598-022-22433-4. PMID 36266435